CLINICAL TRIAL: NCT03038230
Title: A Phase 1, Multinational Study of MCLA-117 in Acute Myelogenous Leukemia
Brief Title: MCLA-117 in Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: strategic considerations
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-117-CL01; 2015-003704-23 (EudraCT Number)
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Myelogenous Leukemia; Acute Myeloid Leukemia
Keywords: human bispecific full length IgG antibody, CLEC12A, CD3; MCLA-117; First in Human; Antibodies, Bispecific; Immunologic Factors; relapsed, refractory patient; AML, minimal residual disease (MRD); Acute Myelogenous Leukemia; Acute Myeloid Leukemia; CD34+CD38; T-cell recruiting
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Neoplasm, Residual | interventions — CD3 Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MCLA-117 bispecific antibody (Experimental): Dose escalation cohorts, with escalating doses of MCLA-117 until MTD or RP2D is reached. The dose is given weekly after initial ramp-up dosing steps. Each Cycle is 28 days. Single agent treatment.
  Part 2-Expansion Cohort: The RP2D of MCLA-117 is given weekly after initial ramp-up dosing steps. Each Cycle is 28 days. Single agent treatment.
  Interventions: Drug: MCLA-117 bispecific antibody

INTERVENTIONS:
Drug: MCLA-117 bispecific antibody — MCLA-117, a human bispecific IgG antibody which targets CLEC12A and CD3
  Other Names: bispecific; human bispecific common light chain; bispecific IgG1 targeting CLEC12A and CD3

SUMMARY:
This is a First-in-Human, single arm, open-label, multi-national study designed to determine the safety, tolerability and preliminary efficacy of MCLA 117.

DETAILED DESCRIPTION:
Study Design :

This open label, single arm, multinational, first-in-human study consists of 2 parts. Part 1 consists of dose escalation cohorts and Part 2 is a dose expansion cohort.

The study population will include adult AML patients (and all subtypes of AML, except for APL) with relapse or refractory disease and newly diagnosed elderly untreated AML patients with high risk cytogenetics. In addition, very high-risk MDS patients with relapsed or refractory disease are eligible.

In Part 1, dose escalations cohorts are followed until dose-limiting toxicity (DLT) or a maximum tolerated dose (MTD) or RecommendedPart2Dose (RP2D) is defined. Dose escalation decisions will be made by the Data Review Committee and will be primarily guided by safety data observed through the end of Cycle 1, as well as on-going assessment of safety beyond Cycle 1 in later cohorts.

Part 2 will begin once the MTD or RP2D is determined in Part 1. Part 2 will further characterize the safety, tolerability, Pharmacokinetic (PK), Pharmacodynamic (PD), immunogenicity and to assess preliminary efficacy of MCLA-117. This part will enroll approximately 30 evaluable patients (defined as evaluable for first efficacy assessment).

For both parts, the study consists of 3 periods: a Screening period (up to 28 days prior to the first dose of study drug); a Treatment period (first dose of study drug until the last dose of study drug with treatment cycles of 28 days); and a Follow Up period (through 30 days after the last dose and quarterly checks for survival data for up to 1 year). Participants' safety will be monitored throughout the study. Patients will be permitted to receive MCLA-117 beyond Cycle 1 if conditions allow this.

Number of Sites:

Approximately 15 centers in five countries are estimated to be involved during Parts 1 and 2 of the study. Additional sites may be added to ensure there is an acceptable enrollment rate or to replace non-enrolling/withdrawn sites.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥18 years old;
2. Signed informed consent form
3. One of the two following:

   i) AML either de novo or secondary [any subtype except acute promyelocytic leukemia (APL)] who either:
   1. are in relapse to standard therapy following an initial response
   2. failed primary induction therapy with no CR (failed ≥2 courses of intensive induction therapy. Intensive chemotherapy defined as an intensity of ≥ 5+2)
   3. newly diagnosed untreated AML in patients ≥ 65 years of age with high risk cytogenetics, if they are not candidates for standard available induction chemotherapy
   4. AML secondary to MDS, either relapsed or refractory, previously treated with hypomethylating agents for at least 4 cycles;
   5. Relapsed or refractory AML unfit for intensive chemotherapy previously treated with a low intensity regimen (e.g. low dose Ara-c, hypomethylating agent, etc.) including Venetoclax for at least 2 cycles;

   OR ii) MDS patients who meet the following criteria: very high-risk disease (IPSS-R score > 6, Greenberg et al., 2012), either relapsed or refractory, previously treated with hypomethylating agents for at least 4 cycles;
4. Must have baseline BM sample taken by BMA/BMB within 28 days prior to first dose of MCLA-117 for CLEC12A detection;
5. Estimated life expectancy of at least 8 weeks;
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
7. Significant toxicities incurred as a result of previous anti-cancer therapy resolved to ≤ Grade 1 (NCI-CTCAE version 4.03);
8. Acceptable laboratory values at screening;
9. Male patients must agree to use an adequate and medically accepted method of contraception throughout the study and for at least 6 months after if their sexual partners are women of child bearing potential (WOCBP).
10. WOCBP must be using highly effective and medically accepted method of contraception to avoid pregnancy throughout the study and for at least 6 months after the study ;
11. WOCBP must have a negative serum or urine pregnancy test within 72 hours prior to the start of study drug.
12. Peripheral blast count </= 30,000/mm3 at the time of initiation of infusion on Cycle 1 Day 1.
13. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. Diagnosis of chronic myelogenous leukemia in blast crisis;
2. Prior hematopoietic stem cell transplantation (this exclusion applies for dose escalation Part 1 and Cohort A of Part 2);
3. For patients in Cohort B of Part 2, prior hematopoietic stem cell transplantation is allowed under certain circumstances.
4. Treatment with anticancer medications, investigational drugs or radiotherapy is allowed within 2 weeks or 5 half-lives prior to start of MCLA-117;
5. Previous receipt of live vaccines in the 4 weeks prior to study drug administration;
6. Chronic concurrent need of use of corticosteroids > 10 mg/day of oral prednisone or the equivalent, except topical preparations (e.g., topical creams, steroid inhaler, nasal spray or ophthalmic solution);
7. Use of immunosuppressant medications within 4 weeks of MCLA-117 administration;
8. Clinically active central nervous system (CNS) leukemia;
9. Patients who are pregnant or lactating;
10. Patients with an active infection or with an unexplained fever during screening or on the first scheduled day of dosing;
11. Patients with known hypersensitivity to any of the components of MCLA-117 or who have had prior hypersensitivity reactions to human or humanized monoclonal antibodies;
12. Patients with known HIV, hepatitis B or C;
13. Patients with New York Heart Association Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50%, or significant uncontrolled cardiac disease, current diagnosis of unstable angina, uncontrolled congestive heart failure, new myocardial infarction, or ventricular arrhythmia requiring medication;
14. Prior malignancy (other than basal cell carcinoma and cervical in situ carcinoma) unless treated with a curative intend and without evidence of malignant disease for 1 year before screening. Patients with prior hematologic malignancies that have progressed to AML (such as Myelodysplastic syndrome, myeloproliferative neoplasms, bi-phenotypic leukemias, AcuteLymphocyticLeukemia) or AML that has relapsed are eligible;
15. Urinary protein >2+ possibly indicative of renal disease. If the 24 hours urine protein shows a result of < 100 mg protein, subject can be eligible;
16. Patients with any other medical or psychological condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results;
17. WOCBP or males with a WOCB partners not willing to use highly effective and medically accepted methods of contraception for 6 months after last study drug administration.
18. Need for concurrent other cytoreductive chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLT) | 28 days
  Evaluation of number of participants with treatment related toxicity observed during a dose escalation step for 1 Cycle

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] | Day 22 predose, 5 minutes prior to End of Infusion (EOI), 1h, 2h, 4h, 8h, 24h, 72h, 6 days after EOI
  Maximum plasma concentration [Cmax] as measured from all individual plasma concentrations
Clearance of plasma | Day 22 predose, 5 minutes prior to End of Infusion (EOI), 1h, 2h, 4h, 8h, 24h, 72h, 6 days after EOI
  Clearance of plasma
Volume of distribution at steady state [Vss] | Day 22 predose, 5 minutes prior to End of Infusion (EOI), 1h, 2h, 4h, 8h, 24h, 72h, 6 days after EOI
  Volume of distribution at steady state [Vss]
Time to reach maximum plasma concentration [Tmax] | Day 22 predose, 5 minutes prior to End of Infusion (EOI), 1h, 2h, 4h, 8h, 24h, 72h, 6 days after EOI
  Time to reach maximum plasma concentration [Tmax]
Half-life [t1/2] | Day 22 predose, 5 minutes prior to End of Infusion (EOI), 1h, 2h, 4h, 8h, 24h, 72h, 6 days after EOI
  Half-life [t1/2] calculated as time from all individual plasma concentrations to reach 50% of maximum concentration
Area under the concentration versus time curve from time zero to time t [AUC0-t] | 1 week
  Area under the concentration versus time curve [AUC0-t]
Incidence of AntiDrugAntibodies (ADA) against MCLA-117 | 24 months
  Number of participants with ADAs against MCLA-117 as measured in serum
Serum titer of ADAs against MCLA-117 | Day 1 of each cycle
  Serum titer of ADAs against MCLA-117 as measured in serum
Serum titer of ADAs against MCLA-117 | Day 28 of each cycle
  Serum titer of ADAs against MCLA-117 as measured in serum
Cytokine levels | Cycle 1: Day 1, 4, 8 and 28 at predose, 4h and 24h after end of infusion
  Change in profile of cytokine upon administration of MCLA-117 compared to baseline
Number of myeloblasts | Day 1 of every cycle and through study completion, an average of 2 months
  number of blasts in peripheral blood and in bone marrow
Objective response | Day 1 of every cycle and through study completion, an average of 2 months
  Objective response is assessed by Cheson 2003

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, PhD, Principal Investigator — Independent Protocol Advisor
Locations (9):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- Ziekenhuis Netwerk Antwerpen Campus Stuivenberg, Antwerp, Belgium
- Institut Gustave Roussy, Villejuif, Île-de-France Region, France
- Fondazione Policlinico Tor Vergata, Rome, Italy
- Netherlands (3):
  - Amsterdam UMC, location VUmc, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No